CLINICAL TRIAL: NCT02511678
Title: Multicenter Study of Cryoablation for Palliation of Painful Bone Metastases
Acronym: MOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGC15-BNE098
Record Dates: First submitted 2015-07-27; First posted 2015-07-30 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Pain; Neoplasm Metastasis; Bone Metastasis of Diverse Origins
MeSH Terms: conditions — Pain; Neoplasm Metastasis | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryoablation (Experimental): All participants will have one cryoablation procedure on one painful metastatic lesion involving bone using a Galil Medical cryoablation system and needles within 14 days of screening. In the case of participants with multiple metastatic lesions involving bone, the most painful lesion is to be selected for cryoablation. If treatment could not be completed within 14 days of screening, the participant will be re-screened using the inclusion and exclusion criteria. Participant preparation, anesthesia, intra-operative monitoring, and postoperative management for the study cryoablation procedure will be identical to those for standard cryoablation treatment routinely performed at the clinical centers that participated in this study and will be at the discretion of the Investigators.
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — The application of repeated freeze and thaw cycles to the identified tissues.
  Other Names: Cryotherapy; Cryosurgery; Visual-ICE™ Cryoablation System; IceSeed® Cryoablation Needle; IceSphere™ Cryoablation Needle; IceRod® PLUS Cryoablation Needle; IceEDGE® 2.4 Cryoablation Needle; IceFORCE® 2.1 Cryoablation Needle; IcePearl® 2.1 Cryoablation Needle

SUMMARY:
This study will evaluate the efficacy of cryoablation for palliation of painful metastases in participants with metastatic lesions involving bone who have failed, are not candidates for, or are not experiencing adequate pain relief from current pain therapies (for example, radiation, analgesics).

DETAILED DESCRIPTION:
Participants with painful metastatic lesions involving bone who meet the eligibility criteria and who have been determined to be an appropriate candidate for cryoablation therapy were offered enrollment into the study. Participants agreeing to participate will read and sign an informed consent form and thus become participants in the study. Treatment will be performed using a Galil Medical cryoablation system and Galil Medical cryoablation needles. Participants will have one cryoablation procedure and will be followed for up to 6 months for palliation of pain, quality of life, and analgesic usage. Baseline and follow-up data will be collected for each participant via a web-based electronic data collection tool.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Metastatic disease involving bone with metastatic disease previously confirmed by prior biopsy; or Metastatic disease involving bone previously confirmed on imaging (for example, computed tomography [CT] or magnetic resonance imaging [MRI]) with known (biopsied) primary disease (primary bone cancer is excluded)
* Current analgesic therapies have failed, the participant is not a candidate for, or the participant is not experiencing adequate pain relief from current pain therapies (for example, radiation, analgesics)
* The 'worst pain' in the last 24 hours must be reported to be 4 or above on a scale of 0 (no pain) to 10 (pain as bad as participant can imagine)
* Pain must be from one painful metastatic lesion involving the bone that is amenable to cryoablation with CT (additional less painful metastatic sites may be present)
* Cryoablation should be performed within 14 days of screening visit
* If taking hormonal therapy, use should be stable (no changes within 4 weeks prior to the cryoablation procedure)
* Karnofsky Performance Scale (KPS) score ≥60
* Life expectancy ≥3 months
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up
* Known coagulopathy or bleeding disorders are controlled

Exclusion Criteria:

* Primary cancer is leukemia, lymphoma, or myeloma
* Tumor involves a weight-bearing long bone of the lower extremity with the tumor causing >50% loss of cortical bone
* Has undergone prior surgery at the tumor site or the index tumor has undergone previous surgery or ablation treatment
* Prior radiation therapy of the index tumor <3 weeks prior to the screening visit
* Index tumor causing clinical or radiographic evidence of spinal cord or cauda equina compression/effacement
* Anticipated treatment of the index tumor that would require iceball formation within 0.5 centimeters (cm) of the spinal cord, brain, other critical nerve structure, or large abdominal vessel (possibly achieved with additional maneuvers such as hydrodissection)
* Index tumor involves the skull
* Currently pregnant, nursing, or wishing to become pregnant during the study
* Serious medical illness, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, or cerebrovascular event within 6 months prior to the screening visit
* Concurrent participation in other studies that could affect the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Jennings, MD, Principal Investigator — Washington University Saint Louis
Locations (11):
- United States (7):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Crittenton Hospital, Rochester, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Rhode Island Hospital, Providence, Rhode Island
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - University Hospital of Strasbourg, Strasbourg
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldfarb HA. Nd:YAG laser laparoscopic coagulation of symptomatic myomas. J Reprod Med. 1992 Jul;37(7):636-8. PMID 1387912
- [Background] Phillips DR, Milim SJ, Nathanson HG, Haselkorn JS. Experience with laparoscopic leiomyoma coagulation and concomitant operative hysteroscopy. J Am Assoc Gynecol Laparosc. 1997 Aug;4(4):425-33. doi: 10.1016/s1074-3804(05)80034-9. PMID 9224575
- [Background] Goldfarb HA. Laparoscopic coagulation of myoma (myolysis). Obstet Gynecol Clin North Am. 1995 Dec;22(4):807-19. No abstract available. PMID 8786884
- [Background] COOPER IS, LEE AS. Cryostatic congelation: a system for producing a limited, controlled region of cooling or freezing of biologic tissues. J Nerv Ment Dis. 1961 Sep;133:259-63. No abstract available. PMID 13881139
- [Background] Saliken JC, Donnelly BJ, Rewcastle JC. The evolution and state of modern technology for prostate cryosurgery. Urology. 2002 Aug;60(2 Suppl 1):26-33. doi: 10.1016/s0090-4295(02)01681-3. PMID 12206845
- [Background] Rewcastle JC, Sandison GA, Saliken JC, Donnelly BJ, McKinnon JG. Considerations during clinical operation of two commercially available cryomachines. J Surg Oncol. 1999 Jun;71(2):106-11. doi: 10.1002/(sici)1096-9098(199906)71:23.0.co;2-z. PMID 10389867
- [Background] Rewcastle JC, Hahn LJ, Saliken JC, McKinnon JG. Use of a moratorium to achieve consistent liquid nitrogen cryoprobe performance. J Surg Oncol. 1997 Oct;66(2):110-3. doi: 10.1002/(sici)1096-9098(199710)66:23.0.co;2-g. PMID 9354166
- [Background] Gage AA. Current progress in cryosurgery. Cryobiology. 1988 Oct;25(5):483-6. doi: 10.1016/0011-2240(88)90056-9. PMID 3197439
- [Background] Gage AA, Guest K, Montes M, Caruana JA, Whalen DA Jr. Effect of varying freezing and thawing rates in experimental cryosurgery. Cryobiology. 1985 Apr;22(2):175-82. doi: 10.1016/0011-2240(85)90172-5. PMID 3979086
- [Background] Gage AA. Progress in cryosurgery. Cryobiology. 1992 Apr;29(2):300-4. doi: 10.1016/0011-2240(92)90030-6. PMID 1582235
- [Background] Homasson JP, Thiery JP, Angebault M, Ovtracht L, Maiwand O. The operation and efficacy of cryosurgical, nitrous oxide-driven cryoprobe. I. Cryoprobe physical characteristics: their effects on cell cryodestruction. Cryobiology. 1994 Jun;31(3):290-304. doi: 10.1006/cryo.1994.1035. PMID 8050273
- [Background] Hamilton A, Hu J. An electronic cryoprobe for cryosurgery using heat pipes and thermoelectric coolers: a preliminary report. J Med Eng Technol. 1993 May-Jun;17(3):104-9. doi: 10.3109/03091909309016215. PMID 8263903
- [Background] Rabin Y, Julian TB, Wolmark N. A compact cryosurgical apparatus for minimally invasive procedures. Biomed Instrum Technol. 1997 May-Jun;31(3):251-8. PMID 9181244
- [Background] Rabin Y, Coleman R, Mordohovich D, Ber R, Shitzer A. A new cryosurgical device for controlled freezing. Cryobiology. 1996 Feb;33(1):93-105. doi: 10.1006/cryo.1996.0010. PMID 8812089
- [Background] Rand RW, Rand RP, Eggerding FA, Field M, Denbesten L, King W, Camici S. Cryolumpectomy for breast cancer: an experimental study. Cryobiology. 1985 Aug;22(4):307-18. doi: 10.1016/0011-2240(85)90178-6. PMID 2992882
- [Background] Miller RH, Mazur P. Survival of frozen-thawed human red cells as a function of cooling and warming velocities. Cryobiology. 1976 Aug;13(4):404-14. doi: 10.1016/0011-2240(76)90096-1. PMID 971585
- [Background] Gage AA, Baust JM, Baust JG. Experimental cryosurgery investigations in vivo. Cryobiology. 2009 Dec;59(3):229-43. doi: 10.1016/j.cryobiol.2009.10.001. Epub 2009 Oct 13. PMID 19833119
- [Background] McTaggart RA, Dupuy DE. Thermal ablation of lung tumors. Tech Vasc Interv Radiol. 2007 Jun;10(2):102-13. doi: 10.1053/j.tvir.2007.09.004. PMID 18070688
- [Background] Callstrom MR, Charboneau JW. Image-guided palliation of painful metastases using percutaneous ablation. Tech Vasc Interv Radiol. 2007 Jun;10(2):120-31. doi: 10.1053/j.tvir.2007.09.003. PMID 18070690
- [Background] McQuay HJ, Collins SL, Carroll D, Moore RA. Radiotherapy for the palliation of painful bone metastases. Cochrane Database Syst Rev. 2000;(2):CD001793. doi: 10.1002/14651858.CD001793. PMID 10796822
- [Background] Callstrom MR, Atwell TD, Charboneau JW, Farrell MA, Goetz MP, Rubin J, Sloan JA, Novotny PJ, Welch TJ, Maus TP, Wong GY, Brown KJ. Painful metastases involving bone: percutaneous image-guided cryoablation--prospective trial interim analysis. Radiology. 2006 Nov;241(2):572-80. doi: 10.1148/radiol.2412051247. PMID 17057075
- [Background] Coleman RE. Management of bone metastases. Oncologist. 2000;5(6):463-70. doi: 10.1634/theoncologist.5-6-463. PMID 11110597
- [Background] Goetz MP, Callstrom MR, Charboneau JW, Farrell MA, Maus TP, Welch TJ, Wong GY, Sloan JA, Novotny PJ, Petersen IA, Beres RA, Regge D, Capanna R, Saker MB, Gronemeyer DH, Gevargez A, Ahrar K, Choti MA, de Baere TJ, Rubin J. Percutaneous image-guided radiofrequency ablation of painful metastases involving bone: a multicenter study. J Clin Oncol. 2004 Jan 15;22(2):300-6. doi: 10.1200/JCO.2004.03.097. PMID 14722039
- [Background] Callstrom MR, Charboneau JW, Goetz MP, Rubin J, Wong GY, Sloan JA, Novotny PJ, Lewis BD, Welch TJ, Farrell MA, Maus TP, Lee RA, Reading CC, Petersen IA, Pickett DD. Painful metastases involving bone: feasibility of percutaneous CT- and US-guided radio-frequency ablation. Radiology. 2002 Jul;224(1):87-97. doi: 10.1148/radiol.2241011613. PMID 12091666
- [Background] Belfiore G, Tedeschi E, Ronza FM, Belfiore MP, Della Volpe T, Zeppetella G, Rotondo A. Radiofrequency ablation of bone metastases induces long-lasting palliation in patients with untreatable cancer. Singapore Med J. 2008 Jul;49(7):565-70. PMID 18695866
- [Background] Hurwitz MD, Ghanouni P, Kanaev SV, Iozeffi D, Gianfelice D, Fennessy FM, Kuten A, Meyer JE, LeBlang SD, Roberts A, Choi J, Larner JM, Napoli A, Turkevich VG, Inbar Y, Tempany CM, Pfeffer RM. Magnetic resonance-guided focused ultrasound for patients with painful bone metastases: phase III trial results. J Natl Cancer Inst. 2014 Apr 23;106(5):dju082. doi: 10.1093/jnci/dju082. PMID 24760791
- [Background] Simon CJ, Dupuy DE. Percutaneous minimally invasive therapies in the treatment of bone tumors: thermal ablation. Semin Musculoskelet Radiol. 2006 Jun;10(2):137-44. doi: 10.1055/s-2006-939031. Epub 2006 Apr 5. PMID 16598666
- [Background] Ullrick SR, Hebert JJ, Davis KW. Cryoablation in the musculoskeletal system. Curr Probl Diagn Radiol. 2008 Jan-Feb;37(1):39-48. doi: 10.1067/j.cpradiol.2007.05.001. PMID 18054665
- [Background] Maiwand MO. The role of cryosurgery in palliation of tracheo-bronchial carcinoma. Eur J Cardiothorac Surg. 1999 Jun;15(6):764-8. doi: 10.1016/s1010-7940(99)00121-9. PMID 10431856
- [Background] Maiwand MO, Homasson JP. Cryotherapy for tracheobronchial disorders. Clin Chest Med. 1995 Sep;16(3):427-43. PMID 8521698
- [Background] Sanderson DR, Neel HB 3rd, Fontana RS. Bronchoscopic cryotherapy. Ann Otol Rhinol Laryngol. 1981 Jul-Aug;90(4 Pt 1):354-8. doi: 10.1177/000348948109000414. PMID 6791555
- [Background] Cozzi PJ, Lynch WJ, Collins S, Vonthethoff L, Morris DL. Renal cryotherapy in a sheep model; a feasibility study. J Urol. 1997 Feb;157(2):710-2. PMID 8996403
- [Background] Gage AA, Fazekas G, Riley EE Jr. Freezing injury to large blood vessels in dogs. With comments on the effect of experimental freezing of bile ducts. Surgery. 1967 May;61(5):748-54. No abstract available. PMID 6024400
- [Background] Gage AM, Montes M, Gage AA. Freezing the canine thoracic aorta in situ. J Surg Res. 1979 Nov;27(5):331-40. doi: 10.1016/0022-4804(79)90149-5. No abstract available. PMID 513700
- [Background] Ladd AP, Rescorla FJ, Baust JG, Callahan M, Davis M, Grosfeld JL. Cryosurgical effects on growing vessels. Am Surg. 1999 Jul;65(7):677-82. PMID 10399979
- [Background] Mandeville AF, McCabe BF. Some observations on the cryobiology of blood vessels. Laryngoscope. 1967 Aug;77(8):1328-50. doi: 10.1288/00005537-196708000-00009. No abstract available. PMID 6034857
- [Background] Callstrom MR, Dupuy DE, Solomon SB, Beres RA, Littrup PJ, Davis KW, Paz-Fumagalli R, Hoffman C, Atwell TD, Charboneau JW, Schmit GD, Goetz MP, Rubin J, Brown KJ, Novotny PJ, Sloan JA. Percutaneous image-guided cryoablation of painful metastases involving bone: multicenter trial. Cancer. 2013 Mar 1;119(5):1033-41. doi: 10.1002/cncr.27793. Epub 2012 Oct 12. PMID 23065947
- [Background] Cleeland CS. The measurement of pain from metastatic bone disease: capturing the patient's experience. Clin Cancer Res. 2006 Oct 15;12(20 Pt 2):6236s-6242s. doi: 10.1158/1078-0432.CCR-06-0988. PMID 17062707
- [Derived] Jennings JW, Prologo JD, Garnon J, Gangi A, Buy X, Palussiere J, Kurup AN, Callstrom M, Genshaft S, Abtin F, Huang AJ, Iannuccilli J, Pilleul F, Mastier C, Littrup PJ, de Baere T, Deschamps F. Cryoablation for Palliation of Painful Bone Metastases: The MOTION Multicenter Study. Radiol Imaging Cancer. 2021 Feb 12;3(2):e200101. doi: 10.1148/rycan.2021200101. eCollection 2021 Mar. PMID 33817650

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Discontinuation reasons reported below of death, withdrew consent, oncologist cancelled study cryoablation, required radiofrequency ablation, negative biopsy, protocol violation, and received radiation treatment include 7 enrolled participants who were discontinued before treatment was attempted. No other data is reported for these 7 participants.
Groups:
- Cryoablation: All participants had one cryoablation procedure on one painful metastatic lesion involving bone using a Galil Medical cryoablation system and needles within 14 days of screening. In the case of participants with multiple metastatic lesions involving bone, the most painful lesion was selected for cryoablation. If treatment could not be completed within 14 days of screening, the participant was re-screened using the inclusion and exclusion criteria. Participant preparation, anesthesia, intra-operative monitoring, and postoperative management for the study cryoablation procedure were identical to those for standard cryoablation treatment routinely performed at the clinical centers that participated in this study and were at the discretion of the Investigators.
Period: Overall Study
Arm/Group | Cryoablation
Started | 73
Intent-to-Treat (ITT) Population | 66 (Participants for whom cryoablation via Galil Medical cryoablation system was attempted or performed.)
Participants Discontinued Pre-Treatment | 7
Safety Population | 65 (Participants for whom received the complete study cryoablation procedure.)
Completed | 37
Not Completed | 36
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 4
Not completed — Death | 19
Not completed — Adverse Event | 1
Not completed — Targeted Therapy to Index Tumor Required | 5
Not completed — Oncologist Cancelled Study Cryoablation | 1
Not completed — Required Radiofrequency Ablation | 1
Not completed — Biopsy was Negative | 1
Not completed — Protocol Violation | 1
Not completed — Received Radiation Treatment | 1

BASELINE CHARACTERISTICS:
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population).
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 27
  More than one race | 0
  Unknown or Not Reported | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Worst Pain Scores as Assessed by the Brief Pain Inventory-Short Form (BPI-SF) at Week 8
Description: The BPI-SF is a validated instrument used widely in clinical research to assess cancer pain. Assessments were of self-reported worst pain scores in the last 24 hours in the target lesion treated with study cryoablation on a scale from 0 (no pain) to 10 (worst pain imaginable) using the BPI-SF. Improvement in self-reported pain scores is defined by ≥2-point reduction in worst pain. A mean difference of a 2-point reduction is considered clinically significant, that is improvement. Baseline data and change from Baseline data at Week 8 is presented.
Time Frame: Baseline, Week 8
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population). The Markov chain Monte Carlo (MCMC) method of imputation was used for imputation of missing BPI-SF values with 50 imputations to be performed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
score on a scale
  Baseline | 7.26 (0.251)
  Change at Week 8 | -2.61 (0.425)
Statistical Analysis 1: Comparison: Cryoablation; Test type: Superiority; p = 0.0746, t-test, 1 sided — The 1-sided p-value was based on a t-test against a performance goal of -2

2. Other Pre Specified Outcome: Percentage of Participants Who Respond to the Cryoablation Therapy
Description: Response was defined as a ≥2-point reduction from baseline in worst pain in last 24 hours with stable medication use (that is, no more than a 25% increase in Morphine Equivalent Daily Dose [MEDD] from baseline). MEDD is calculated using the following formula: [Dose]*[MEDD Factor]. MEDD Factor is based on the type and dose of the opioid received. Pain was assessed using BPI-SF with a scale of 0 (no pain) to 10 (worst pain imaginable). Percentages are proportion of responders based on logistic regression after MCMC, multiple imputation. For visits where medication use is not available, morphine equivalent values from the most recent non-missing visit are used.
Time Frame: Baseline and Week 8
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
percentage of participants | 42.1 [29.9 to 55.4]

3. Other Pre Specified Outcome: Change From Baseline in QoL as Indicated by the Overall Average BPI-SF Interference Score at Weeks 1, 4, 8, 12, 16, 20, and 24.
Description: Quality of Life (QoL) as indicated by the change in overall average BPI-SF Pain Interference score from baseline to each visit was evaluated at Weeks 1, 4, 8, 12, 16, 20, and 24. Using the BPI-SF, participants rated the amount of interference from pain on a scale of 0 (does not interfere) to 10 (completely interferes) for the following areas: general activity. mood, walking ability, relations, sleep, and enjoyment. For participants with responses ≥50% of the areas at a time point, a total Pain Interference score, which was the mean of the individual area scores, was calculated programmatically at that point. Baseline data and change from Baseline data is presented.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable interference from pain scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 65
score on a scale
  General Activity, Baseline | 6.6 (2.9)
  General Activity, Change at Week 1: number analyzed (Participants) | 64
  General Activity, Change at Week 1 | -1.6 (3.8)
  General Activity, Change at Week 4: number analyzed (Participants) | 53
  General Activity, Change at Week 4 | -2.2 (3.9)
  General Activity, Change at Week 8: number analyzed (Participants) | 50
  General Activity, Change at Week 8 | -2.4 (4.0)
  General Activity, Change at Week 12: number analyzed (Participants) | 40
  General Activity, Change at Week 12 | -2.9 (3.9)
  General Activity, Change at Week 16: number analyzed (Participants) | 35
  General Activity, Change at Week 16 | -3.3 (4.0)
  General Activity, Change at Week 20: number analyzed (Participants) | 32
  General Activity, Change at Week 20 | -2.7 (4.6)
  General Activity, Change at Week 24: number analyzed (Participants) | 32
  General Activity, Change at Week 24 | -3.4 (3.5)
  Mood, Baseline | 5.1 (2.9)
  Mood, Change at Week 1: number analyzed (Participants) | 64
  Mood, Change at Week 1 | -1.3 (3.4)
  Mood, Change at Week 4: number analyzed (Participants) | 53
  Mood, Change at Week 4 | -2.0 (3.7)
  Mood, Change at Week 8: number analyzed (Participants) | 49
  Mood, Change at Week 8 | -2.4 (3.1)
  Mood, Change at Week 12: number analyzed (Participants) | 39
  Mood, Change at Week 12 | -2.7 (3.1)
  Mood, Change at Week 16: number analyzed (Participants) | 36
  Mood, Change at Week 16 | -2.7 (3.5)
  Mood, Change at Week 20: number analyzed (Participants) | 33
  Mood, Change at Week 20 | -2.4 (3.9)
  Mood, Change at Week 24: number analyzed (Participants) | 33
  Mood, Change at Week 24 | -2.6 (3.4)
  Walking Ability, Baseline | 5.7 (3.4)
  Walking Ability, Change at Week 1: number analyzed (Participants) | 64
  Walking Ability, Change at Week 1 | -1.7 (3.4)
  Walking Ability, Change at Week 4: number analyzed (Participants) | 53
  Walking Ability, Change at Week 4 | -1.8 (3.5)
  Walking Ability, Change at Week 8: number analyzed (Participants) | 49
  Walking Ability, Change at Week 8 | -1.4 (3.4)
  Walking Ability, Change at Week 12: number analyzed (Participants) | 39
  Walking Ability, Change at Week 12 | -1.9 (3.5)
  Walking Ability, Change at Week 16: number analyzed (Participants) | 35
  Walking Ability, Change at Week 16 | -2.5 (3.3)
  Walking Ability, Change at Week 20: number analyzed (Participants) | 32
  Walking Ability, Change at Week 20 | -2.3 (3.51)
  Walking Ability, Change at Week 24: number analyzed (Participants) | 32
  Walking Ability, Change at Week 24 | -2.3 (2.9)
  Normal Work, Baseline: number analyzed (Participants) | 64
  Normal Work, Baseline | 6.4 (3.2)
  Normal Work, Change at Week 1: number analyzed (Participants) | 62
  Normal Work, Change at Week 1 | -1.2 (3.5)
  Normal Work, Change at Week 4: number analyzed (Participants) | 51
  Normal Work, Change at Week 4 | -2.6 (4.1)
  Normal Work, Change at Week 8: number analyzed (Participants) | 49
  Normal Work, Change at Week 8 | -2.1 (4.0)
  Normal Work, Change at Week 12: number analyzed (Participants) | 40
  Normal Work, Change at Week 12 | -2.5 (4.6)
  Normal Work, Change at Week 16: number analyzed (Participants) | 35
  Normal Work, Change at Week 16 | -3.2 (4.4)
  Normal Week, Change at Week 20: number analyzed (Participants) | 32
  Normal Week, Change at Week 20 | -2.5 (4.6)
  Normal Week, Change at Week 24: number analyzed (Participants) | 32
  Normal Week, Change at Week 24 | -3.0 (3.7)
  Relations, Baseline | 4.0 (3.1)
  Relations, Change at Week 1: number analyzed (Participants) | 64
  Relations, Change at Week 1 | -1.8 (3.2)
  Relations, Change at Week 4: number analyzed (Participants) | 53
  Relations, Change at Week 4 | -1.7 (3.7)
  Relations, Change at Week 8: number analyzed (Participants) | 50
  Relations, Change at Week 8 | -1.5 (3.2)
  Relations, Change at Week 12: number analyzed (Participants) | 40
  Relations, Change at Week 12 | -2.2 (3.2)
  Relations, Change at Week 16: number analyzed (Participants) | 36
  Relations, Change at Week 16 | -2.4 (3.3)
  Relations, Change at Week 20: number analyzed (Participants) | 33
  Relations, Change at Week 20 | -2.5 (3.8)
  Relations, Change at Week 24: number analyzed (Participants) | 33
  Relations, Change at Week 24 | -2.4 (3.1)
  Sleep, Baseline | 5.8 (3.2)
  Sleep, Change at Week 1: number analyzed (Participants) | 64
  Sleep, Change at Week 1 | -2.2 (3.1)
  Sleep, Change at Week 4: number analyzed (Participants) | 53
  Sleep, Change at Week 4 | -2.5 (3.8)
  Sleep, Change at Week 8: number analyzed (Participants) | 50
  Sleep, Change at Week 8 | -2.3 (3.3)
  Sleep, Change at Week 12: number analyzed (Participants) | 40
  Sleep, Change at Week 12 | -3.1 (3.2)
  Sleep, Change at Week 16: number analyzed (Participants) | 36
  Sleep, Change at Week 16 | -4.1 (3.4)
  Sleep, Change at Week 20: number analyzed (Participants) | 33
  Sleep, Change at Week 20 | -2.5 (3.9)
  Sleep, Change at Week 24: number analyzed (Participants) | 33
  Sleep, Change at Week 24 | -3.0 (3.9)
  Enjoyment, Baseline | 5.4 (3.6)
  Enjoyment, Change at Week 1: number analyzed (Participants) | 63
  Enjoyment, Change at Week 1 | -1.9 (3.4)
  Enjoyment, Change at Week 4: number analyzed (Participants) | 52
  Enjoyment, Change at Week 4 | -2.5 (3.5)
  Enjoyment, Change at Week 8: number analyzed (Participants) | 50
  Enjoyment, Change at Week 8 | -2.2 (3.4)
  Enjoyment, Change at Week 12: number analyzed (Participants) | 40
  Enjoyment, Change at Week 12 | -2.8 (3.1)
  Enjoyment, Change at Week 16: number analyzed (Participants) | 36
  Enjoyment, Change at Week 16 | -3.4 (3.5)
  Enjoyment, Change at Week 20: number analyzed (Participants) | 33
  Enjoyment, Change at Week 20 | -2.6 (4.3)
  Enjoyment, Change at Week 24: number analyzed (Participants) | 32
  Enjoyment, Change at Week 24 | -3.3 (3.2)
  Total Pain, Baseline | 5.5 (2.5)
  Total Pain, Change at Week 1: number analyzed (Participants) | 64
  Total Pain, Change at Week 1 | -1.7 (2.6)
  Total Pain, Change at Week 4: number analyzed (Participants) | 53
  Total Pain, Change at Week 4 | -2.2 (3.1)
  Total Pain, Change at Week 8: number analyzed (Participants) | 50
  Total Pain, Change at Week 8 | -2.0 (2.8)
  Total Pain, Change at Week 12: number analyzed (Participants) | 40
  Total Pain, Change at Week 12 | -2.6 (2.8)
  Total Pain, Change at Week 16: number analyzed (Participants) | 36
  Total Pain, Change at Week 16 | -3.1 (2.8)
  Total Pain, Change at Week 20: number analyzed (Participants) | 33
  Total Pain, Change at Week 20 | -2.5 (3.2)
  Total Pain, Change at Week 24: number analyzed (Participants) | 33
  Total Pain, Change at Week 24 | -2.9 (2.3)

4. Other Pre Specified Outcome: Change From Baseline in Physical Function as Assessed by the KPS Scale at Weeks 1, 4, 8, 12, 16, 20, and 24
Description: The Karnofsky Performance Status (KPS) scale is a standard way of measuring the ability of cancer participants to perform ordinary tasks. KPS may be used to determine a participant's prognosis and to measure changes in a participant's ability to function. Assessments made by examining the change in the baseline scores to those reported post-operatively. KPS scores range from 0 to 100. A higher score means the participant is better able to carry out daily activities from Baseline to 1, 4, 8, 12, 16, 20, and 24 weeks after cryoablation. Baseline data and change from Baseline data is presented.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable KPS scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
units on a scale
  Baseline | 80.6 (14.5)
  Change at Week 1: number analyzed (Participants) | 64
  Change at Week 1 | -5.0 (10.8)
  Change at Week 4: number analyzed (Participants) | 56
  Change at Week 4 | -4.5 (11.4)
  Change at Week 8: number analyzed (Participants) | 52
  Change at Week 8 | -7.3 (15.7)
  Change at Week 12: number analyzed (Participants) | 41
  Change at Week 12 | -5.4 (14.3)
  Change at Week 16: number analyzed (Participants) | 39
  Change at Week 16 | -3.6 (14.1)
  Change at Week 20: number analyzed (Participants) | 37
  Change at Week 20 | -7.0 (16.0)
  Change at Week 24: number analyzed (Participants) | 36
  Change at Week 24 | -7.5 (18.4)

5. Other Pre Specified Outcome: Number of Participants With Additional Pain Therapies
Description: Participants requiring additional targeted therapies to the index tumor (for example, cryoablation, radio frequency ablation [RFA], microwave ablation [MWA], high intensity focused ultrasound [HIFU], radiation, surgery) were withdrawn from the study. Other therapies, including pain medication and chemotherapy, were permitted during the study. All additional therapies were recorded. The number of participants requiring new therapy since the last visit is presented.
Time Frame: Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable additional pain therapy data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
Participants
  Week 1: number analyzed (Participants) | 64
  Week 1 | 17
  Week 4: number analyzed (Participants) | 58
  Week 4 | 30
  Week 8: number analyzed (Participants) | 52
  Week 8 | 29
  Week 12: number analyzed (Participants) | 41
  Week 12 | 24
  Week 16: number analyzed (Participants) | 39
  Week 16 | 25
  Week 20: number analyzed (Participants) | 37
  Week 20 | 21
  Week 24: number analyzed (Participants) | 37
  Week 24 | 18

6. Other Pre Specified Outcome: Change From Baseline in MEDD and NSAID Doses at Weeks 1, 4, 8, 12, 16, 20, and 24
Description: Analgesic (that is, opioid or non-steroidal anti-inflammatory drug [NSAID]) use and the reason for each change in analgesic dose was recorded at each study visit. Opioid medications were converted to a standardized MEDD. MEDD is calculated using the following formula: [Dose]*[MEDD Factor]. MEDD Factor is based on the type and dose of the opioid received. Baseline data and change from Baseline data is presented.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable MEDD and NSAID data.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
milligrams (mg)
  MEDD, Baseline | 31.365 (69.9231)
  MEDD, Change at Week 1: number analyzed (Participants) | 64
  MEDD, Change at Week 1 | 4.123 (44.0061)
  MEDD, Change at Week 4: number analyzed (Participants) | 57
  MEDD, Change at Week 4 | 5.884 (55.6215)
  MEDD, Change at Week 8: number analyzed (Participants) | 51
  MEDD, Change at Week 8 | -0.466 (37.1101)
  MEDD, Change at Week 12: number analyzed (Participants) | 41
  MEDD, Change at Week 12 | 2.019 (41.4507)
  MEDD, Change at Week 16: number analyzed (Participants) | 39
  MEDD, Change at Week 16 | 7.404 (20.9301)
  MEDD, Change at Week 20: number analyzed (Participants) | 37
  MEDD, Change at Week 20 | 8.927 (20.2095)
  MEDD, Change at Week 24: number analyzed (Participants) | 37
  MEDD, Change at Week 24 | 4.392 (15.0878)
  NSAID, Baseline: number analyzed (Participants) | 65
  NSAID, Baseline | 60.8 (251.32)
  NSAID, Change at Week 1: number analyzed (Participants) | 64
  NSAID, Change at Week 1 | 4.1 (126.15)
  NSAID, Change at Week 4: number analyzed (Participants) | 57
  NSAID, Change at Week 4 | -6.1 (278.40)
  NSAID, Change at Week 8: number analyzed (Participants) | 51
  NSAID, Change at Week 8 | -6.1 (371.14)
  NSAID, Change at Week 12: number analyzed (Participants) | 41
  NSAID, Change at Week 12 | -32.9 (401.50)
  NSAID, Change at Week 16: number analyzed (Participants) | 39
  NSAID, Change at Week 16 | -53.8 (342.47)
  NSAID, Change at Week 20: number analyzed (Participants) | 37
  NSAID, Change at Week 20 | -55.4 (304.09)
  NSAID, Change at Week 24: number analyzed (Participants) | 37
  NSAID, Change at Week 24 | -68.9 (312.55)

7. Other Pre Specified Outcome: Change From Baseline in Worst Pain Scores as Assessed by the BPI-SF at Weeks 1, 4, 12, 16, 20, and 24
Description: The BPI-SF is a validated instrument used widely in clinical research to assess cancer pain. Assessments were of self-reported worst pain scores in the last 24 hours in the target lesion treated with study cryoablation on a scale from 0 (no pain) to 10 (worst pain imaginable) using the BPI-SF. Improvement in self-reported pain scores is defined by ≥2-point reduction in worst pain. A mean difference of a 2 point reduction is considered clinically significant, that is improvement. Baseline data and change from Baseline data at Weeks 1, 4, 12, 16, 20, and 24 is presented.
Time Frame: Baseline, Week 1, Week 4, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable worse pain scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 66
score on a scale
  Baseline | 7.3 (2.04)
  Change at Week 1: number analyzed (Participants) | 64
  Change at Week 1 | -2.0 (2.6)
  Change at Week 4: number analyzed (Participants) | 54
  Change at Week 4 | -2.6 (3.12)
  Change at Week 8: number analyzed (Participants) | 50
  Change at Week 8 | -2.5 (3.23)
  Change at Week 12: number analyzed (Participants) | 40
  Change at Week 12 | -3.3 (3.53)
  Change at Week 16: number analyzed (Participants) | 37
  Change at Week 16 | -3.6 (3.46)
  Change at Week 20: number analyzed (Participants) | 34
  Change at Week 20 | -3.5 (3.32)
  Change at Week 24: number analyzed (Participants) | 34
  Change at Week 24 | -3.4 (3.22)

8. Other Pre Specified Outcome: Change From Baseline in Average Pain Scores as Assessed by the BPI-SF at Weeks 1, 4, 8, 12, 16, 20, and 24
Description: The BPI-SF is a validated instrument used widely in clinical research to assess cancer pain. Assessments were of self-reported average pain scores in the last 24 hours in the target lesion treated with study cryoablation on a scale from 0 (no pain) to 10 (worst pain imaginable) using the BPI-SF. Baseline data and change from Baseline data is presented.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable average pain scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryoablation
Number analyzed (Participants) | 65
score on a scale
  Baseline | 5.6 (1.93)
  Change at Week 1: number analyzed (Participants) | 64
  Change at Week 1 | -1.6 (2.49)
  Change at Week 4: number analyzed (Participants) | 53
  Change at Week 4 | -2.1 (2.65)
  Change at Week 8: number analyzed (Participants) | 50
  Change at Week 8 | -1.8 (2.66)
  Change at Week 12: number analyzed (Participants) | 40
  Change at Week 12 | -2.6 (2.5)
  Change at Week 16: number analyzed (Participants) | 37
  Change at Week 16 | -2.8 (2.73)
  Change at Week 20: number analyzed (Participants) | 34
  Change at Week 20 | -2.4 (2.75)
  Change at Week 24: number analyzed (Participants) | 34
  Change at Week 24 | -2.8 (2.48)

9. Other Pre Specified Outcome: Self-Assessed Overall Treatment Effect (OTE) at Weeks 1, 4, 8, 12, 16, 20, and 24
Description: Participants performed a self-assessment of OTE at Week 1 and every visit thereafter (Weeks 4, 8, 12, 16, 20 and 24). Participants were asked their opinion of the effect cryoablation procedure had on their wellbeing and asked to compare their wellbeing at the time of each follow-up visit to the previous visit or phone call. The wellbeing categories were "Better than the Last Visit," "The Same as the Last Visit," and "Worse than the Last Visit." The percentage of participants that were reported for each wellbeing category at Weeks 1, 4, 8, 12, 16, 20, and 24 is presented.
Time Frame: Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: Participants for whom cryoablation via a Galil Medical cryoablation system was attempted or performed (ITT Population) and evaluable OTE data.
Measure: Number; unit: percentage of participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 64
percentage of participants
  Better than the Last Visit, Week 1 | 60.9
  Better than the Last Visit, Week 4: number analyzed (Participants) | 58
  Better than the Last Visit, Week 4 | 58.6
  Better than the Last Visit, Week 8: number analyzed (Participants) | 52
  Better than the Last Visit, Week 8 | 48.1
  Better than the Last Visit, Week 12: number analyzed (Participants) | 41
  Better than the Last Visit, Week 12 | 39.0
  Better than the Last Visit, Week 16: number analyzed (Participants) | 39
  Better than the Last Visit, Week 16 | 38.5
  Better than the Last Visit, Week 20: number analyzed (Participants) | 37
  Better than the Last Visit, Week 20 | 27.0
  Better than the Last Visit, Week 24: number analyzed (Participants) | 37
  Better than the Last Visit, Week 24 | 29.7
  Same as the Last Visit, Week 1 | 26.6
  Same as the Last Visit, Week 4: number analyzed (Participants) | 58
  Same as the Last Visit, Week 4 | 24.1
  Same as the Last Visit, Week 8: number analyzed (Participants) | 52
  Same as the Last Visit, Week 8 | 36.5
  Same as the Last Visit, Week 12: number analyzed (Participants) | 41
  Same as the Last Visit, Week 12 | 51.2
  Same as the Last Visit, Week 16: number analyzed (Participants) | 39
  Same as the Last Visit, Week 16 | 48.7
  Same as the Last Visit, Week 20: number analyzed (Participants) | 37
  Same as the Last Visit, Week 20 | 56.8
  Same as the Last Visit, Week 24: number analyzed (Participants) | 37
  Same as the Last Visit, Week 24 | 56.8
  Worse than the Last Visit, Week 1 | 12.5
  Worse than the Last Visit, Week 4: number analyzed (Participants) | 58
  Worse than the Last Visit, Week 4 | 12.1
  Worse than the Last Visit, Week 8: number analyzed (Participants) | 52
  Worse than the Last Visit, Week 8 | 13.5
  Worse than the Last Visit, Week 12: number analyzed (Participants) | 41
  Worse than the Last Visit, Week 12 | 9.8
  Worse than the Last Visit, Week 16: number analyzed (Participants) | 39
  Worse than the Last Visit, Week 16 | 12.8
  Worse than the Last Visit, Week 20: number analyzed (Participants) | 37
  Worse than the Last Visit, Week 20 | 13.5
  Worse than the Last Visit, Week 24: number analyzed (Participants) | 37
  Worse than the Last Visit, Week 24 | 10.8
  Missing, Week 1 | 0
  Missing, Week 4: number analyzed (Participants) | 58
  Missing, Week 4 | 5.2
  Missing, Week 8: number analyzed (Participants) | 52
  Missing, Week 8 | 1.9
  Missing, Week 12: number analyzed (Participants) | 41
  Missing, Week 12 | 0
  Missing, Week 16: number analyzed (Participants) | 39
  Missing, Week 16 | 0
  Missing, Week 20: number analyzed (Participants) | 37
  Missing, Week 20 | 2.7
  Missing, Week 24: number analyzed (Participants) | 37
  Missing, Week 24 | 2.7

10. Other Pre Specified Outcome: Number of Participants With Intra- or Post-operative Adverse Events, a Serious Adverse Event, or Unanticipated Adverse Device Effects
Description: The number of participants with an intra-operative non-serious adverse event, a post-operative, a non-serious adverse event, a serious adverse event, or unanticipated adverse device effects related to the cryoablation procedure is presented. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to 30 days post-cryoablation
Population: Participants for whom received the complete study cryoablation procedure (Safety Population).
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 65
Participants
  Intra-operative non-serious adverse event | 3
  Post-operative non-serious adverse event | 3
  Non-serious event after discharge within 30 days | 8
  Serious adverse event | 3
  Unanticipated adverse device effect | 0

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: All-Cause Mortality reported for all Enrolled Participants. Adverse Events were monitored and reported for participants who received the complete study cryoablation procedure (Safety Population [N=65]).
Arm/Group | Cryoablation
All-Cause Mortality (participants affected / at risk) | 19/73
Serious Adverse Events (participants affected / at risk) | 3/65
Other Adverse Events (participants affected / at risk) | 13/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation (N=65)
Abdominal pain (Gastrointestinal disorders) | 1
Burn (Injury, poisoning and procedural complications) | 1
Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cryoablation (N=65)
Pericardial Effusion (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Localized Edema (General disorders) | 1
Pain at needle site (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neuralgia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Galil Medical can require Investigator to postpone publications/presentations for up to 12 months so data from all sites can be published. Galil Medical will limit review of Investigator's draft to confirm Confidential Information is not being disclosed. If Galil Medical notes publishing Study results may affect obtaining a patent, Investigator may not publish for up to 60 days until patent application is filed. Investigator will acknowledge Galil Medical in any publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT02511678/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT02511678/SAP_001.pdf